CLINICAL TRIAL: NCT02974855
Title: A MULTICENTER, OPEN-LABEL, MULTIPLE ASCENDING DOSE STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS, AND EFFICACY OF SUBCUTANEOUS OR INTRAVENOUS PF-06741086 IN SUBJECTS WITH SEVERE HEMOPHILIA
Brief Title: PF-06741086 Multiple Dose Study in Severe Hemophilia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: B7841002; 2016-001885-27 (EudraCT Number)
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Hemophilia A or B
Keywords: hemophilia
MeSH Terms: conditions — Hemophilia A | interventions — marstacimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF-06741086 (Cohort 1) (Experimental)
  Interventions: Biological: PF-06741086
- PF-06741086 (Cohort 2) (Experimental)
  Interventions: Biological: PF-06741086
- PF-06741086 (Cohort 3) (Experimental)
  Interventions: Biological: PF-06741086
- PF-06741086 (Cohort 4) (Experimental)
  Interventions: Biological: PF-06741086

INTERVENTIONS:
Biological: PF-06741086 — PF-06741086 subcutaneous (SC) injection
  Arms: PF-06741086 (Cohort 1)
Biological: PF-06741086 — PF-06741086 SC injection
  Arms: PF-06741086 (Cohort 2)
Biological: PF-06741086 — PF-06741086 SC injection
  Arms: PF-06741086 (Cohort 3)
Biological: PF-06741086 — PF-06741086 SC injection
  Arms: PF-06741086 (Cohort 4)

SUMMARY:
This study is designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of multiple subcutaneous and/or intravenous doses of PF-06741086 in subjects with severe hemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Severe hemophilia A or B (Factor VIII or Factor IX activity ≤ 1%), including patients with inhibitors to Factor VIII or Factor IX
* Episodic (on-demand) treatment regimen prior to screening
* At least 6 acute bleeding episodes during the 6-month period prior to screening

Exclusion Criteria:

* Known coronary artery, thrombotic, or ischemic disease
* Currently receiving treatment for acute bleeding episodes with APCC and cannot substitute treatment with rFVIIa

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 27 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (4):
  - UC Denver Hemophilia and Thrombosis Center - Pharmacy, Aurora, Colorado
  - UC Denver Hemophilia and Thrombosis Center, Aurora, Colorado
  - Pharmacy, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
- Hospital Dr. Sotero del Rio, Santiago, Chile
- Klinicki bolnicki centar Zagreb, Zagreb, Croatia
- Klinika Hematologii i Transplantologii Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
- South Africa (2):
  - Phoenix Pharma (Pty) Ltd, Port Elizabeth, Eastern Cape
  - Haemophilia Comprehensive Care Centre, Johannesburg, Gauteng
- UniversitatsSpital Zurich, Klinik fur Hamatologie, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Mahlangu JN, Lamas JL, Morales JC, Malan DR, Salek SZ, Wang M, Boggio LN, Hegemann I, Mital A, Cardinal M, Zhu T, Sun P, Arkin S. A phase 1b/2 clinical study of marstacimab, targeting human tissue factor pathway inhibitor, in haemophilia. Br J Haematol. 2023 Jan;200(2):229-239. doi: 10.1111/bjh.18420. Epub 2022 Aug 23. PMID 35999026
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7841002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 27 participants were enrolled in the study and assigned to 1 of 4 cohorts. Only 26 participants received the study treatment and 1 participant withdrew after randomization but prior to dosing.
Groups:
- PF-06741086 300 mg SC QW Non-Inhibitor: Participants without inhibitors to Factor VIII (FVIII) or Factor IX (FIX) in this cohort received PF-06741086 300 mg subcutaneously (SC) once weekly (QW) from Day 1 to Day 78.
- PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor: Participants without inhibitors to Factor VIII (FVIII) or Factor IX (FIX) in this cohort received PF-06741086 300 mg loading dose on Day 1 and 150 mg subcutaneously (SC) once weekly (QW) from Day 8 to Day 78.
- PF-06741086 450 mg SC QW Non-Inhibitor: Participants without inhibitors to Factor VIII (FVIII) or Factor IX (FIX) in this cohort received PF-06741086 450 mg subcutaneously (SC) once weekly (QW) from Day 1 to Day 78.
- PF-06741086 300 mg SC QW Inhibitor: Participants with inhibitors to Factor VIII (FVIII) or Factor IX (FIX) in this cohort received PF-06741086 300 mg subcutaneously (SC) once weekly (QW) from Day 1 to Day 78.
Period: Overall Study
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor
Started | 7 | 6 | 6 | 7
Completed | 7 | 5 | 6 | 6
Not Completed | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 6 | 7 | 26
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.9 (8.17) | 28.7 (8.31) | 41.7 (15.87) | 44.1 (9.44) | 36.7 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 6 | 6 | 7 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 0 | 4 | 12
  White | 3 | 2 | 6 | 3 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect. AEs included both SAEs and non-serious AEs. TEAEs were AEs occurred following the start of treatment or AEs increasing in severity during treatment. Severe TEAEs were TEAEs that interfered significantly with participants' usual function. Treatment-related TEAEs were determined by the investigator.
Time Frame: Study Day 1 to Day 113 Visit
Population: The analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Overall PF-06741086 300 mg SC: The overall PF-06741086 300 mg SC group combined participants from both the PF-06741086 300 mg SC QW non-inhibitor and inhibitor dose cohorts.
- Total: The total group combined participants from all PF-06741086 cohorts in this study.
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Participants
  All-causalities TEAE | 7 | 4 | 6 | 4 | 11 | 21
  Treatment-related TEAE | 4 | 4 | 3 | 3 | 7 | 14
  All-causalities serious TEAE | 1 | 1 | 1 | 1 | 2 | 4
  Treatment-related serious TEAE | 0 | 0 | 0 | 0 | 0 | 0
  All-causalities Grade 3 or 4 TEAE | 0 | 0 | 2 | 2 | 2 | 4
  Treatment-related Grade 3 or 4 TEAE | 0 | 0 | 2 | 2 | 2 | 4

2. Primary Outcome: Number of Participants Discontinued From Study Due to TEAEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment. TEAEs were AEs occurred following the start of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator.
Time Frame: Study Day 1 to Day 113 Visit
Population: The analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Participants
  All-causalities TEAE | 0 | 1 | 0 | 1 | 1 | 2
  Treatment-related TEAE | 0 | 1 | 0 | 1 | 1 | 2

3. Primary Outcome: Number of Participants With Abnormal Laboratory Findings-Hematology
Description: Hematology evaluation included: hemoglobin, hematocrit, erythrocytes, platelets, leukocytes, lymphocytes, neutrophils, basophils, eosinophils and monocytes. Predefined criteria for hemoglobin and hematocrit: <0.8*lower limit of normal (LLN) or <0.8*Baseline(Baseline <1.0*LLN); for platelets: <100,000*10^3/mm^3 or <= 0.77*Baseline (Baseline <1.0*LLN).
Time Frame: Baseline to Study Day 113 Visit
Population: This analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Participants
  Hemoglobin meeting pre-defined criteria | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit meeting pre-defined criteria | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes <0.8*LLN | 0 | 0 | 0 | 0 | 0 | 0
  Platelets meeting pre-defined criteria | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes <0.6*LLN | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes >1.5*upper limit of normal (ULN) | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes <0.8*LLN | 0 | 1 | 0 | 0 | 0 | 1
  Lymphocytes >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils <0.8*LLN | 1 | 2 | 0 | 0 | 1 | 3
  Neutrophils >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Basophils >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Laboratory Findings-Clinical Chemistry
Description: Clinical chemistry evaluation included bilirubin, direct and indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, alkaline phosphatase, protein, albumin, urea nitrogen, creatinine, urate, triglycerides, sodium, potassium, chloride, calcium, bicarbonate, glucose, creatine kinase, troponin I, cholesterol and fibrinogen.
Time Frame: Baseline to Study Day 113
Population: This analysis population included all participants who received at least 1 dose of investigational product. Number analyzed refers to number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Participants
  Bilirubin >1.5*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Direct Bilirubin >1.5*ULN: number analyzed (Participants) | 0 | 3 | 1 | 0 | 0 | 4
  Direct Bilirubin >1.5*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Indirect Bilirubin >1.5*ULN: number analyzed (Participants) | 0 | 3 | 1 | 0 | 0 | 4
  Indirect Bilirubin >1.5*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase >3.0*ULN | 0 | 0 | 1 | 0 | 0 | 1
  Alanine Aminotransferase >3.0*ULN | 1 | 1 | 1 | 0 | 1 | 3
  Gamma Glutamyl Transferase >3.0*ULN: number analyzed (Participants) | 0 | 3 | 1 | 0 | 0 | 4
  Gamma Glutamyl Transferase >3.0*ULN | 0 | 1 | 0 | 0 | 0 | 1
  Alkaline Phosphatase | 0 | 0 | 0 | 0 | 0 | 0
  Protein <0.8*LLN | 0 | 0 | 0 | 0 | 0 | 0
  Protein >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Albumin <0.8*LLN | 0 | 0 | 0 | 0 | 0 | 0
  Albumin >1.2*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen >1.3*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine >1.3*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Urate >1.2*ULN | 0 | 0 | 0 | 2 | 2 | 2
  Triglycerides >1.3*ULN: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  Triglycerides >1.3*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Sodium <0.95*LLN | 0 | 0 | 0 | 0 | 0 | 0
  Sodium >1.05*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Potassium <0.9*LLN | 1 | 0 | 0 | 0 | 1 | 1
  Potassium >1.1*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Chloride <0.9*LLN | 0 | 0 | 0 | 0 | 0 | 0
  Chloride >1.1*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Calcium <0.9*LLN | 0 | 0 | 0 | 0 | 0 | 0
  Calcium >1.1*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Bicarbonate <0.9*LLN | 2 | 1 | 0 | 0 | 2 | 3
  Bicarbonate >1.1*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Glucose <0.6*LLN | 0 | 0 | 0 | 0 | 0 | 0
  Glucose >1.5*ULN | 0 | 0 | 2 | 1 | 1 | 3
  Creatine Kinase >2.0*ULN: number analyzed (Participants) | 0 | 3 | 1 | 0 | 0 | 26
  Creatine Kinase >2.0*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Troponin I >1.0*ULN | 1 | 1 | 0 | 2 | 3 | 4
  Cholesterol >1.3*ULN: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 1
  Cholesterol >1.3*ULN | 0 | 0 | 0 | 0 | 0 | 0
  Fibrinogen <=0.5*LLN or <=0.5*baseline | 0 | 0 | 0 | 1 | 1 | 1

5. Primary Outcome: Number of Participants With Abnormal Laboratory Findings-Urinalysis
Description: Urinalysis included: pH, urine glucose, ketones, urine protein, urine hemoglobin, urobilinogen, urine bilirubin, nitrite, leukocyte esterase, urine erythrocytes, urine leukocytes and bacteria.
Time Frame: Baseline to Study Day 113 Visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Participants
  pH (Scalar) <4.5 | 0 | 0 | 0 | 0 | 0 | 0
  pH (Scalar) >8 | 0 | 0 | 0 | 0 | 0 | 0
  Urine glucose >=1 | 0 | 0 | 1 | 0 | 0 | 1
  Ketones (Scalar) >=1 | 0 | 0 | 1 | 1 | 1 | 2
  Urine protein >=1 | 0 | 0 | 0 | 1 | 1 | 1
  Urine hemoglobin (Scalar) >=1 | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen >=1 | 0 | 0 | 0 | 0 | 0 | 0
  Urine bilirubin (Scalar) >=1 | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite (Scalar) >=1 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte esterase (Scalar) >=1 | 1 | 1 | 0 | 1 | 2 | 3
  Urine erythrocytes (/HPF) >=20: number analyzed (Participants) | 1 | 0 | 0 | 2 | 3 | 3
  Urine erythrocytes (/HPF) >=20 | 0 | 0 | 0 | 0 | 0 | 0
  Urine leukocytes (/HPF) >=20: number analyzed (Participants) | 1 | 1 | 0 | 3 | 4 | 5
  Urine leukocytes (/HPF) >=20 | 0 | 1 | 0 | 1 | 1 | 2
  Bacteria (/HPF) >20: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 2
  Bacteria (/HPF) >20 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Change From Baseline for Globulin by Dose Cohort
Description: Blood samples were obtained to determine globulin level in serum, total globulin was derived as total protein other than albumin.
Time Frame: Baseline, Study Day 8, 15, 22, 29, 57, 85 and 113.
Population: This analysis population included all participants randomized and who had received at least 1 dose of randomized treatment. Number analyzed refers to number of participants evaluable for specified rows of time points.
Measure: Mean (Standard Deviation); unit: gram/liter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
gram/liter
  Globulin, Change at Day 8 | -0.3 (3.04) | -1.7 (3.93) | -1.3 (2.73) | 0.4 (2.51) | 0.1 (2.70) | -0.7 (3.01)
  Globulin, Change at Day 15 | -0.7 (2.06) | -0.8 (2.32) | -1.3 (2.50) | -1.3 (3.35) | -1.0 (2.69) | -1.0 (2.47)
  Globulin, Study Day 22 | -1.6 (2.82) | -0.5 (1.52) | -1.5 (3.08) | -0.6 (4.12) | -1.1 (3.43) | -1.0 (2.93)
  Globulin, Change at Day 29: number analyzed (Participants) | 6 | 6 | 5 | 7 | 13 | 24
  Globulin, Change at Day 29 | -0.3 (3.27) | -0.3 (3.08) | 0.2 (1.10) | -1.3 (2.75) | -0.8 (2.91) | -0.5 (2.62)
  Globulin, Change at Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 24
  Globulin, Change at Day 57 | 0.7 (3.72) | 1.8 (2.99) | -0.3 (1.63) | -0.7 (2.94) | 0.0 (3.28) | 0.4 (2.90)
  Globulin, Change at Day 85: number analyzed (Participants) | 7 | 5 | 6 | 6 | 13 | 24
  Globulin, Change at Day 85 | 1.3 (3.15) | -1.4 (4.77) | -0.5 (3.02) | 1.0 (2.61) | 1.2 (2.79) | 0.2 (3.35)
  Globulin, Change at Day 113: number analyzed (Participants) | 7 | 6 | 4 | 6 | 13 | 23
  Globulin, Change at Day 113 | -0.3 (3.15) | -1.2 (4.67) | 0.5 (2.65) | -0.8 (3.06) | -0.5 (2.99) | -0.5 (3.33)

7. Primary Outcome: Change From Baseline for Prothrombin International Normalized Ratio (PT/INR) by Dose Cohort
Description: Blood samples were obtained to evaluate this ratio. The prothrombin time (PT) is a test that helps evaluate your ability to appropriately form blood clots. The international normalized ratio (INR) is a calculation based on results of a PT that is used to monitor individuals who are being treated with the blood-thinning medication (anticoagulant) warfarin (Coumadin®).
Time Frame: Baseline, Study Day 8, 15, 22, 29, 57, 85 and 113.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Ratio
  PT/INR, Change at Day 8 | -0.03 (0.049) | -0.02 (0.041) | 0.05 (0.138) | 0.03 (0.138) | 0.00 (0.104) | 0.01 (0.102)
  PT/INR, Change at Day 15 | 0.03 (0.076) | 0.00 (0.063) | 0.02 (0.041) | 0.00 (0.082) | 0.01 (0.077) | 0.01 (0.065)
  PT/INR, Change at Day 22 | 0.03 (0.095) | 0.00 (0.063) | -0.02 (0.041) | -0.01 (0.069) | 0.01 (0.083) | 0.00 (0.069)
  PT/INR, Change at Day 29: number analyzed (Participants) | 6 | 6 | 6 | 7 | 13 | 25
  PT/INR, Change at Day 29 | 0.03 (0.082) | -0.02 (0.041) | 0.00 (0.063) | 0.00 (0.115) | 0.02 (0.099) | 0.00 (0.079)
  PT/INR, Change at Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 24
  PT/INR, Change at Day 57 | 0.00 (0.126) | -0.03 (0.052) | 0.00 (0.063) | -0.02 (0.075) | -0.01 (0.100) | -0.01 (0.080)
  PT/INR, Change at Day 85: number analyzed (Participants) | 7 | 5 | 6 | 6 | 13 | 24
  PT/INR, Change at Day 85 | -0.01 (0.107) | 0.04 (0.152) | -0.02 (0.075) | -0.03 (0.082) | -0.02 (0.093) | -0.01 (0.102)
  PT/INR, Change at Day 113: number analyzed (Participants) | 7 | 6 | 4 | 6 | 13 | 23
  PT/INR, Change at Day 113 | 0.06 (0.127) | -0.03 (0.052) | -0.05 (0.058) | 0.07 (0.052) | 0.06 (0.096) | 0.02 (0.094)

8. Primary Outcome: Change From Baseline for Activated Partial Thromboplastin Time (aPTT) by Dose Cohort
Description: The activated partial thromboplastin time (aPTT) is a screening test that helps evaluate a person's ability to appropriately form blood clots. It measures the number of seconds it takes for a clot to form in a sample of blood after substances (reagents) are added. Blood sample were obtained to evaluate aPTT.
Time Frame: Baseline, Study Day 8, 15, 22, 29, 57, 85 and 113.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
seconds
  aPTT, Change at Day 8 | 8.49 (17.017) | 10.63 (11.634) | 11.03 (15.467) | -12.26 (7.082) | -1.89 (16.512) | 3.98 (16.079)
  aPTT, Change at Day 15 | 9.50 (10.907) | 12.50 (15.303) | 1.20 (20.075) | -10.26 (6.757) | -0.38 (13.457) | 2.96 (15.825)
  aPTT, Change at Day 22 | 14.79 (10.799) | 12.15 (15.232) | 4.50 (9.765) | -11.77 (11.247) | 1.51 (17.381) | 4.65 (15.543)
  aPTT, Change at Day 29: number analyzed (Participants) | 6 | 6 | 6 | 7 | 13 | 25
  aPTT, Change at Day 29 | 13.42 (11.102) | 9.85 (15.999) | 10.13 (10.250) | -12.87 (11.390) | -0.74 (17.386) | 4.41 (16.009)
  aPTT, Change at Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 24
  aPTT, Change at Day 57 | 13.65 (13.378) | 14.25 (14.061) | 7.82 (11.580) | -9.13 (8.390) | 2.26 (15.966) | 6.65 (14.817)
  aPTT, Change at Day 85: number analyzed (Participants) | 7 | 5 | 6 | 6 | 13 | 24
  aPTT, Change at Day 85 | 9.00 (10.928) | 3.84 (18.089) | 7.68 (14.733) | -7.57 (10.124) | 1.35 (13.278) | 3.45 (14.257)
  aPTT, Change at Day 113: number analyzed (Participants) | 7 | 6 | 4 | 6 | 13 | 23
  aPTT, Change at Day 113 | 8.46 (23.391) | 0.78 (16.332) | -0.97 (26.633) | 9.37 (20.265) | 8.88 (21.093) | 5.05 (20.500)

9. Primary Outcome: Change From Baseline for Fibrinogen by Dose Cohort
Description: Fibrinogen is a protein, specifically a clotting factor (factor I), that is essential for proper blood clot formation. Blood samples were obtained to evaluate the amount of fibrinogen.
Time Frame: Baseline, Study Day 8, 15, 22, 29, 57, 85 and 113.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milligram/deciliter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
milligram/deciliter
  Fibrinogen, Change at Day 8 | -49.7 (28.72) | -59.7 (38.20) | -3.5 (24.16) | -54.4 (59.58) | -52.1 (45.00) | -42.6 (44.14)
  Fibrinogen, Change at Day 15 | -59.4 (41.28) | -51.0 (31.84) | -8.3 (25.96) | -85.6 (94.86) | -72.5 (71.58) | -52.7 (60.78)
  Fibrinogen, Change at Day 22 | -72.0 (40.76) | -36.8 (44.93) | -33.2 (32.41) | -87.9 (115.49) | -79.9 (83.61) | -59.2 (69.08)
  Fibrinogen, Change at Day 29: number analyzed (Participants) | 6 | 6 | 6 | 7 | 13 | 25
  Fibrinogen, Change at Day 29 | -84.7 (43.53) | -40.0 (26.57) | -40.3 (20.99) | -99.9 (106.59) | -92.8 (80.82) | -67.6 (65.01)
  Fibrinogen, Change at Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 24
  Fibrinogen, Change at Day 57 | -33.5 (85.81) | 10.0 (79.34) | -21.3 (24.23) | -58.7 (71.81) | -46.1 (76.57) | -25.9 (69.68)
  Fibrinogen, Change at Day 85: number analyzed (Participants) | 7 | 5 | 6 | 6 | 13 | 24
  Fibrinogen, Change at Day 85 | -49.9 (47.93) | -39.4 (63.27) | -10.5 (44.94) | -40.8 (74.28) | -45.7 (58.91) | -35.6 (56.31)
  Fibrinogen, Change at Day 113: number analyzed (Participants) | 7 | 6 | 4 | 6 | 13 | 23
  Fibrinogen, Change at Day 113 | -38.6 (44.48) | -5.2 (29.34) | 23.5 (26.80) | -61.7 (126.18) | -49.2 (88.13) | -25.1 (73.56)

10. Primary Outcome: Change From Baseline for Antithrombin III by Dose Cohort
Description: Antithrombin (AT) is a protein produced by the liver that helps regulate blood clot formation (i.e., a naturally-occurring mild blood thinner). Blood samples were collected to measure the activity (function) and the amount (quantity) of antithrombin in an individual's blood is used to evaluate the person for excessive blood clotting.
Time Frame: Baseline, Study Day 8, 15, 22 and 29.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of activity of AT in plasma
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Percentage of activity of AT in plasma
  Antithrombin III, Change at Day 8 | 2.1 (5.18) | -1.8 (7.05) | 3.7 (7.58) | -7.3 (9.32) | -2.6 (8.74) | -1.0 (8.24)
  Antithrombin III, Change at Day 15 | 2.4 (16.96) | 0.5 (8.14) | -15.3 (16.45) | -6.9 (6.74) | -2.2 (13.30) | -4.6 (14.02)
  Antithrombin III, Change at Day 22 | -7.6 (17.55) | 5.2 (12.69) | -5.3 (9.97) | -4.4 (17.61) | -6.0 (16.97) | -3.3 (14.97)
  Antithrombin III, Change at Day 29: number analyzed (Participants) | 6 | 6 | 6 | 7 | 13 | 25
  Antithrombin III, Change at Day 29 | -0.8 (8.04) | -4.3 (11.55) | -10.3 (15.45) | -12.7 (12.96) | -7.2 (12.20) | -7.3 (12.51)

11. Primary Outcome: Change From Baseline for Troponin I by Dose Cohort
Description: Blood samples were collected to measure the level of cardiac-specific troponin I in the blood to help detect heart injury.
Time Frame: Baseline, Study Day 8, 15, 22, 29, 57 and 85.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
nanogram/milliliter
  Troponin I, Change at Day 8: number analyzed (Participants) | 7 | 4 | 5 | 5 | 12 | 21
  Troponin I, Change at Day 8 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Troponin I, Change at Day 15: number analyzed (Participants) | 7 | 4 | 5 | 6 | 13 | 22
  Troponin I, Change at Day 15 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Troponin I, Change at Day 22: number analyzed (Participants) | 6 | 4 | 5 | 6 | 12 | 21
  Troponin I, Change at Day 22 | 0.0042 (0.01021) | 0 (0) | 0 (0) | 0.0142 (0.03470) | 0.0092 (0.02494) | 0.0052 (0.01907)
  Troponin I, Change at Day 29: number analyzed (Participants) | 6 | 4 | 5 | 7 | 13 | 22
  Troponin I, Change at Day 29 | 0 (0) | 0.0113 (0.02250) | 0 (0) | 0.0121 (0.03213) | 0.0065 (0.02357) | 0.0059 (0.02010)
  Troponin I, Change at Day 57: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 1
  Troponin I, Change at Day 57 |  | 0 |  |  |  | 0
  Troponin I, Change at Day 85: number analyzed (Participants) | 1 | 0 | 0 | 0 | 1 | 1
  Troponin I, Change at Day 85 | 0 |  |  |  | 0 | 0

12. Primary Outcome: Number of Participants With Vital Signs Data Meeting Pre-specified Criteria
Description: Criteria for potentially clinically important findings in vital signs data were defined as: 1) supine systolic blood pressure (BP): value <90 mm Hg or change >=30 mm Hg increase; 2) Supine diastolic BP: value <50 mm Hg or change >=20 mm Hg increase; 3) Supine pulse rate: value <40 beats/min or >120 beats/min.
Time Frame: Baseline to Study Day 113 Visit
Population: This analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Participants
  Supine systolic BP value <90 mm Hg | 0 | 0 | 0 | 0 | 0 | 0
  Supine systolic BP change >=30 mm Hg increase | 0 | 1 | 1 | 0 | 0 | 2
  Supine diastolic BP value <50 mm Hg | 0 | 0 | 0 | 0 | 0 | 0
  Supine diastolic BP change >=20 mm Hg increase | 0 | 1 | 0 | 0 | 0 | 1
  Supine pulse rate value <40 beats/min | 0 | 0 | 0 | 0 | 0 | 0
  Supine pulse rate value >120 beats/min | 0 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Change Meeting Pre-specified Criteria
Description: Criteria for potentially clinically important changes in ECG were defined as: PR interval baseline >200 msec and increase of >=25%; PR interval baseline <=200 msec and increase of >=50%; QRS interval increase of >=50%. Only the number of participants meeting pre-defined criteria was reported below.
Time Frame: Baseline to Study Day 29 Visit.
Population: This analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Participants | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examination Findings
Description: Physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. Clinical significance was judged by the investigator.
Time Frame: Baseline to Study Day 113 Visit
Population: This analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Participants | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Number of Participants With Infusion and Injection Site Reactions
Description: Infusion and injection site reactions included: injection site bruising, injection site erythema, injection site haemorrhage, injection site induration, injection site pain, injection site pruritus, injection site swelling and injection site warmth. Grade of severity was defined as follows: Mild: Transient or mild discomfort (< 48 hours); no medical intervention/therapy required. Moderate: Mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required. Severe: Marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible.
Time Frame: Baseline to Study Day 113 Visit
Population: This analysis population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Participants
  All-causality Mild | 3 | 1 | 0 | 1 | 4 | 5
  Treatment-related Mild | 3 | 1 | 0 | 1 | 4 | 5
  All-causality Moderate | 0 | 0 | 0 | 1 | 1 | 1
  Treatment-related Moderate | 0 | 0 | 0 | 1 | 1 | 1
  All-causality Severe | 0 | 0 | 2 | 0 | 0 | 2
  Treatment-related Severe | 0 | 0 | 2 | 0 | 0 | 2

16. Secondary Outcome: Annualized Bleeding Rate (ABR)
Description: Pre-treatment ABR = number of bleeding episodes within 6 months prior to study enrollment (total number of bleeding episodes in hemophilia history CRF) × 2; On-study ABR = number of bleeding episodes occurred within 9 days after the last dose / ([last dose date + 9 - first dose date + 1] / 365.25) The historical On Demand group was constructed using the following internal Pfizer studies: ReFacto AF 3082B2-4432 (B1831004), BeneFIX B1821010, and BeneFIX 3090A1-400 (B1821004). Participants who were on On Demand treatment in B1831004, as well as data from the On Demand period in B1821004 and B1821010 were used to construct the historical On Demand group. The resulting dataset were further filtered to match the key inclusion/exclusion criteria of Study B7841002 based on age and factor activity (18 <=age <=65 and factor activity <=1%).
Time Frame: Pre-treatment: within 6 months prior to study enrollment; On-study: Day 1 to 9 days after the last dose (Day 78)
Population: This efficacy analysis was conducted in the Per Protocol Analysis Set (PPAS) that included all participants who received at least 1 dose of investigational product and did not have any major protocol deviations.
Measure: Mean (Standard Deviation); unit: Bleeding episodes per year
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 24
Bleeding episodes per year
  Pre-Treatment | 23.00 (7.457) | 14.67 (1.633) | 20.33 (10.838) | 17.33 (3.011) | 20.17 (6.177) | 18.83 (7.100)
  On-Study | 4.22 (3.799) | 1.62 (2.533) | 4.17 (6.467) | 0.65 (1.603) | 2.43 (3.345) | 2.67 (4.092)
Statistical Analysis 1: Comparison: PF-06741086 300 mg SC QW Non-Inhibitor; The comparator was the Historical on Demand Group; Test type: Superiority — Prophylactic treatment with PF-06741086 will be considered superior to On Demand treatment with respect to ABR reduction if 1) the upper limit of the 2-sided 80%CI of the ratio of ABR in PF/historical On Demand is <1 and 2) the estimate of the ratio of ABR in PF/historical On Demand ≤0.3. Drug will be considered not superior to On Demand treatment if the lower limit of the 2-sided 80%CI of the ratio of PF/historical On Demand >0.3; p = 0.0002, Negative Binomial Model; ratio = 0.15, 80% CI 2-sided [0.08 to 0.29]
Statistical Analysis 2: Comparison: PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor; The comparator was the Historical on Demand Group; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.0001, Negative Binomial Model; ratio = 0.05, 80% CI 2-sided [0.02 to 0.14]
Statistical Analysis 3: Comparison: PF-06741086 450 mg SC QW Non-Inhibitor; The comparator was the Historical on Demand Group; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.0002, Negative Binomial Model; ratio = 0.15, 80% CI 2-sided [0.08 to 0.29]
Statistical Analysis 4: Comparison: PF-06741086 300 mg SC QW Inhibitor; The comparator was the Historical on Demand Group; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.0005, Negative Binomial Model; ratio = 0.03, 80% CI 2-sided [0.01 to 0.10]
Statistical Analysis 5: Comparison: Overall PF-06741086 300 mg SC; The comparator was the Historical on Demand Group; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p < 0.0001, Negative Binomial Model; ratio = 0.09, 80% CI 2-sided [0.05 to 0.16]
Statistical Analysis 6: Comparison: PF-06741086 300 mg SC QW Non-Inhibitor; On-Study versus Pre-Treatment; Test type: Superiority; p < 0.0001, Negative Binomial Model; ratio = 0.18, 80% CI 2-sided [0.11 to 0.31]
Statistical Analysis 7: Comparison: PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor; On-Study versus Pre-Treatment; Test type: Superiority; p = 0.0002, Negative Binomial Model; ratio = 0.10, 80% CI 2-sided [0.04 to 0.22]
Statistical Analysis 8: Comparison: PF-06741086 450 mg SC QW Non-Inhibitor; On-Study versus Pre-Treatment; Test type: Superiority; p = 0.0154, Negative Binomial Model; ratio = 0.20, 80% CI 2-sided [0.09 to 0.47]
Statistical Analysis 9: Comparison: PF-06741086 300 mg SC QW Inhibitor; On-Study versus Pre-Treatment; Test type: Superiority; p = 0.0005, Negative Binomial Model; ratio = 0.04, 80% CI 2-sided [0.01 to 0.14]
Statistical Analysis 10: Comparison: Overall PF-06741086 300 mg SC; On-Study versus Pre-Treatment; Test type: Superiority; p < 0.0001, Negative Binomial Model; ratio = 0.12, 80% CI 2-sided [0.08 to 0.20]

17. Secondary Outcome: Plasma PF-06741086 Concentrations
Description: Plasma PF-06741086 concentrations were analyzed using a validated, sensitive and specific electrochemiluminescence (ECL) method.
Time Frame: pre-dose on Study Day 1, 24hours (h), 72h post Study Day 1 dosing, pre-dose on Study Day 8, 15 and 22, pre-dose on Study Day 29, 24h, 96h post Study Day 29 dosing, pre-dose on Study Day 57, 168h, 840h post Study Day 57 dosing
Population: The PK concentration population included all enrolled participants treated who had at least 1 quantifiable concentration. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
nanogram/milliliter
  Pre-dose on Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
  24h post Day 1 dosing | 12180 (8500.2) | 15620 (8055.3) | 11640 (4670.6) | 18130 (9111.3) | 15150 (9011.0)
  72h post Day 1 dosing | 17560 (10637) | 20850 (8433.7) | 24270 (8018.9) | 20640 (8978.4) | 19100 (9591.3)
  Pre-dose on Day 8 | 11290 (10019) | 14060 (6201.2) | 16700 (5689.1) | 11940 (4981.7) | 11610 (7609.2)
  Pre-dose on Day 15 | 22850 (15142) | 16680 (7668.8) | 28180 (10163) | 24870 (5726.8) | 23860 (11048)
  Pre-dose on Day 22: number analyzed (Participants) | 7 | 6 | 5 | 6 | 13
  Pre-dose on Day 22 | 33010 (19724) | 17900 (10509) | 41200 (17504) | 36450 (10432) | 34600 (15590)
  Pre-dose on Day 29: number analyzed (Participants) | 5 | 6 | 4 | 5 | 10
  Pre-dose on Day 29 | 46180 (21357) | 16780 (7939.7) | 59950 (30625) | 41500 (13884) | 43840 (17161)
  24h post Day 29 dosing: number analyzed (Participants) | 5 | 6 | 4 | 5 | 10
  24h post Day 29 dosing | 66500 (27135) | 23530 (8548.4) | 73780 (22425) | 69920 (27902) | 68210 (26010)
  96h post Day 29 dosing: number analyzed (Participants) | 3 | 4 | 4 | 4 | 7
  96h post Day 29 dosing | 69130 (30459) | 20680 (11580) | 74950 (27538) | 58150 (18753) | 62860 (22794)
  Pre-dose on Day 57: number analyzed (Participants) | 5 | 5 | 6 | 5 | 10
  Pre-dose on Day 57 | 54580 (29022) | 18260 (15062) | 66480 (45529) | 59140 (24377) | 56860 (25382)
  168h post Day 57 dosing: number analyzed (Participants) | 5 | 4 | 5 | 5 | 10
  168h post Day 57 dosing | 53890 (43483) | 24800 (2994.4) | 87500 (37163) | 66700 (28971) | 60300 (35481)
  840h post Day 57 dosing: number analyzed (Participants) | 3 | 0 | 0 | 1 | 4
  840h post Day 57 dosing | 586.6 (1318.4) |  |  | 90.00 (180.00) | 406.0 (1056.1)

18. Secondary Outcome: Area Under the Concentration-time Profile From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of PF-06741086
Description: AUClast was calculated by linear/Log trapezoidal method.
Time Frame: Pre-dose on Day 1, 24 and 96 hours post Day 1 dosing
Population: The PK parameter analysis population included all enrolled participants treated who had at least 1 quantifiable concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
nanogram*hour/milliliter | 1818000 (79) | 2675000 (41) | 2806000 (37) | 2495000 (40) | 2130000 (61)

19. Secondary Outcome: Maximum Plasma Concentration (Cmax) of PF-06741086
Description: Cmax was observed directly from data.
Time Frame: Pre-dose on Day 1, 24 and 96 hours post Day 1 dosing, pre-dose on Day 29, 24 and 96 hours post Day 29 dosing
Population: The PK parameter analysis population included all enrolled participants treated who had at least 1 quantifiable concentration. Number analyzed refers to number of participants evaluable for specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
nanogram/milliliter
  Cmax, Day 1 | 14880 (70) | 19480 (42) | 23070 (37) | 19680 (51) | 17110 (61)
  Cmax, Day 29: number analyzed (Participants) | 5 | 6 | 4 | 5 | 10
  Cmax, Day 29 | 61850 (47) | 24150 (44) | 73490 (38) | 66070 (44) | 63930 (43)

20. Secondary Outcome: Lowest Concentration Observed During the Dosing Interval (Cmin) of PF-06741086
Description: Cmin was observed directly from data.
Time Frame: Pre-dose on Day 1, 24 and 96 hours post Day 1 dosing, pre-dose on Day 29, 24 and 96 hours post Day 29 dosing
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
nanogram/milliliter
  Cmin, Day 1 | 7980 (112) | 13040 (43) | 15660 (44) | 11140 (41) | 9429 (78)
  Cmin, Day 29: number analyzed (Participants) | 5 | 6 | 4 | 5 | 10
  Cmin, Day 29 | 42120 (52) | 15000 (59) | 53630 (61) | 39490 (37) | 40790 (42)

21. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of PF-06741086
Description: Tmax was observed directly from data as time of first occurrence.
Time Frame: Pre-dose on Day 1, 24 and 96 hours post Day 1 dosing, pre-dose on Day 29, 24 and 96 hours post Day 29 dosing
Population: as for outcome 19
Measure: Median (Full Range); unit: hours
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
hours
  Tmax, Day 1 | 70.0 [69.1 to 72.8] | 69.7 [68.2 to 71.1] | 71.6 [67.6 to 72.3] | 70.7 [22.8 to 167] | 70.1 [22.8 to 167]
  Tmax, Day 29: number analyzed (Participants) | 5 | 6 | 4 | 5 | 10
  Tmax, Day 29 | 23.7 [23.1 to 94.2] | 23.7 [22.0 to 71.7] | 58.5 [23.3 to 97.0] | 22.8 [22.1 to 94.7] | 23.3 [22.1 to 94.7]

22. Secondary Outcome: Area Under the Serum Concentration-time Curve Over the Dosing Interval Tau (AUCtau) of PF-06741086
Description: The dosing interval tau was 1 week. AUCtau was obtained by linear/log trapezoidal method.
Time Frame: Pre-dose on Day 29, 24 and 96 hours post Day 29 dosing
Population: The PK parameter analysis population included all enrolled participants treated who had at least 1 quantifiable concentration and in whom at least 1 of the PK parameters of interest was calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
nanogram*hour/milliliter | 9045000 (49) | 3309000 (50) | 11090000 (43) | 9248000 (38) | 9146000 (41)

23. Secondary Outcome: Apparent Clearance After Oral Dose (CL/F) of PF-06741086
Description: CL/F was calculated by dose/AUCtau.
Time Frame: Pre-dose on Day 29, 24 and 96 hours post Day 29 dosing
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter/hour
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
milliliter/hour | 33.16 (49) | 45.34 (50) | 40.60 (43) | 32.43 (38) | 32.79 (41)

24. Secondary Outcome: Change From Baseline in Total Tissue Factor Pathway Inhibitor (TFPI)
Description: Total amount of tissue factor pathway inhibitor (TFPI) (bound and unbound) in plasma. TFPI is a protease inhibitor which acts as an antagonist of the extrinsic coagulation pathway via inhibition of tissue factor activated coagulation factor VII (FVIIa) and activated factor X (FXa). Human plasma samples were analyzed for total TFPI concentrations using a validated, sensitive and specific high-performance liquid chromatography tandem mass spectrometric method (LC-MS/MS). Mixed model repeated measures (MMRM) was used to analyze the change from baseline on TFPI.
Time Frame: Baseline, Study Day 2, 4, 8, 15, 22, 29, 30, 33, 57, 85 and 113
Population: The analysis population included all enrolled participants who received at least 1 dose of study medication and had a baseline measurement and at least 1 post-dose measurement for at least 1 pharmacodynamic endpoint.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
nanogram/milliliter
  TFPI, Change at Day 2: number analyzed (Participants) | 7 | 5 | 6 | 7 | 14
  TFPI, Change at Day 2 | 3.9 (31.43) | -13.4 (17.17) | 8.2 (19.83) | 0.4 (46.81) | 2.1 (38.35)
  TFPI, Change at Day 4: number analyzed (Participants) | 7 | 5 | 6 | 7 | 14
  TFPI, Change at Day 4 | 39.4 (46.10) | 43.2 (25.76) | 74.0 (22.03) | 86.0 (29.71) | 62.7 (44.41)
  TFPI, Change at Day 8: number analyzed (Participants) | 7 | 5 | 6 | 7 | 14
  TFPI, Change at Day 8 | 42.7 (82.52) | 72.4 (10.81) | 120.5 (34.41) | 55.9 (69.84) | 49.3 (73.76)
  TFPI, Change at Day 15: number analyzed (Participants) | 7 | 5 | 6 | 7 | 14
  TFPI, Change at Day 15 | 143.9 (107.56) | 78.8 (43.36) | 186.5 (52.80) | 156.1 (83.87) | 150.0 (92.88)
  TFPI, Change at Day 22: number analyzed (Participants) | 7 | 4 | 6 | 7 | 14
  TFPI, Change at Day 22 | 256.1 (137.09) | 110.0 (80.96) | 301.5 (84.39) | 223.3 (128.08) | 239.7 (128.59)
  TFPI, Change at Day 29: number analyzed (Participants) | 6 | 5 | 6 | 7 | 13
  TFPI, Change at Day 29 | 324.2 (127.46) | 106.6 (77.56) | 334.7 (120.67) | 222.1 (135.29) | 269.2 (136.83)
  TFPI, Change at Day 30: number analyzed (Participants) | 7 | 6 | 5 | 6 | 12
  TFPI, Change at Day 30 | 363.8 (156.87) | 115.6 (86.41) | 347.8 (170.70) | 286.7 (103.72) | 325.3 (133.04)
  TFPI, Change at Day 33: number analyzed (Participants) | 6 | 4 | 5 | 6 | 12
  TFPI, Change at Day 33 | 337.7 (129.05) | 165.8 (35.20) | 351.0 (161.54) | 296.3 (112.30) | 317.0 (117.34)
  TFPI, Change at Day 57: number analyzed (Participants) | 6 | 5 | 6 | 6 | 12
  TFPI, Change at Day 57 | 383.3 (137.17) | 140.0 (126.96) | 460.5 (247.37) | 371.0 (178.73) | 377.2 (152.03)
  TFPI, Change at Day 85: number analyzed (Participants) | 7 | 3 | 6 | 6 | 13
  TFPI, Change at Day 85 | 396.7 (216.54) | 246.7 (51.81) | 492.2 (308.46) | 425.0 (266.57) | 409.8 (230.80)
  TFPI, Change at Day 113: number analyzed (Participants) | 7 | 2 | 4 | 6 | 13
  TFPI, Change at Day 113 | 30.0 (72.30) | 41.5 (28.99) | 39.0 (16.15) | -14.0 (33.17) | 9.7 (59.94)

25. Secondary Outcome: Change From Baseline in Thrombin Generation (TGA) Lag Time
Description: An ex vivo pharmacodynamic measure of thrombin generation (initiation of thrombin generation), the lag time is the time needed to form the first traces of thrombin.
Time Frame: Baseline, Study Day 2, 4, 8, 15, 22, 29, 30, 33, 57, 85 and 113
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
minutes
  TGA lag time, Change at Day 2 | -7.16 (5.865) | -2.77 (1.517) | -3.93 (1.919) | -4.13 (1.238) | -5.64 (4.365)
  TGA lag time, Change at Day 4 | -6.80 (6.079) | -2.80 (1.399) | -3.48 (1.957) | -4.17 (1.501) | -5.49 (4.467)
  TGA lag time, Change at Day 8 | -6.94 (5.882) | -2.88 (1.292) | -3.57 (2.018) | -4.43 (1.506) | -5.69 (4.327)
  TGA lag time, Change at Day 15 | -6.90 (5.897) | -3.07 (1.221) | -3.27 (1.870) | -4.29 (1.342) | -5.59 (4.327)
  TGA lag time, Change at Day 22 | -6.94 (5.978) | -2.80 (1.585) | -3.12 (2.097) | -4.34 (1.638) | -5.64 (4.422)
  TGA lag time, Change at Day 29: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  TGA lag time, Change at Day 29 | -5.33 (4.871) | -2.77 (1.392) | -3.43 (2.016) | -4.32 (1.781) | -4.83 (3.537)
  TGA lag time, Change at Day 30: number analyzed (Participants) | 6 | 6 | 6 | 5 | 11
  TGA lag time, Change at Day 30 | -5.22 (4.893) | -2.77 (1.372) | -3.50 (2.082) | -4.48 (1.681) | -4.88 (3.640)
  TGA lag time, Change at Day 33: number analyzed (Participants) | 6 | 6 | 6 | 5 | 11
  TGA lag time, Change at Day 33 | -5.08 (4.414) | -2.40 (1.568) | -3.35 (2.261) | -4.52 (1.771) | -4.83 (3.329)
  TGA lag time, Change at Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  TGA lag time, Change at Day 57 | -4.73 (4.711) | -2.28 (2.020) | -3.42 (1.962) | -3.78 (1.376) | -4.26 (3.346)
  TGA lag time,Change at Day 85: number analyzed (Participants) | 7 | 5 | 6 | 6 | 13
  TGA lag time,Change at Day 85 | -6.34 (5.745) | -3.10 (1.344) | -3.27 (2.014) | -3.33 (1.755) | -4.95 (4.497)
  TGA lag time, Change at Day 113: number analyzed (Participants) | 7 | 2 | 4 | 6 | 13
  TGA lag time, Change at Day 113 | -0.79 (7.428) | 0.80 (0.283) | 1.53 (5.306) | 0.78 (5.251) | -0.06 (6.304)

26. Secondary Outcome: Change From Baseline in Thrombin Generation (TGA) Peak
Description: An ex vivo pharmacodynamic measure of thrombin generation (initiation of thrombin generation). The peak represents the highest thrombin concentration that can be generated. There may be patients who reach the peak faster or slower than others and this may represent hyper- or hypocoagulability, respectively.
Time Frame: Baseline, Study Day 2, 4, 8, 15, 22, 29, 30, 33, 57, 85 and 113
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: nanomole
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
nanomole
  TGA peak, Change at Day 2 | 72.93 (35.734) | 70.92 (23.721) | 68.18 (15.693) | 63.41 (9.743) | 68.17 (25.642)
  TGA peak, Change at Day 4 | 60.00 (30.196) | 59.28 (30.156) | 50.87 (20.687) | 51.79 (14.929) | 55.89 (23.278)
  TGA peak, Change at Day 8 | 49.36 (32.033) | 56.00 (33.636) | 50.30 (14.019) | 54.36 (15.007) | 51.86 (24.171)
  TGA peak, Change at Day 15 | 49.01 (23.471) | 52.57 (28.440) | 46.40 (22.985) | 40.90 (7.886) | 44.96 (17.340)
  TGA peak, Change at Day 22 | 44.50 (27.260) | 52.07 (33.558) | 38.15 (16.313) | 44.41 (22.567) | 44.46 (24.042)
  TGA peak, Change at Day 29: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  TGA peak, Change at Day 29 | 42.95 (24.026) | 49.72 (29.316) | 38.23 (21.808) | 42.48 (23.057) | 42.72 (22.452)
  TGA peak, Change at Day 30: number analyzed (Participants) | 6 | 6 | 6 | 5 | 11
  TGA peak, Change at Day 30 | 35.93 (26.177) | 51.75 (29.276) | 37.72 (24.136) | 48.62 (21.427) | 41.70 (23.878)
  TGA peak, Change at Day 33: number analyzed (Participants) | 6 | 6 | 6 | 5 | 11
  TGA peak, Change at Day 33 | 76.68 (69.887) | 46.83 (37.084) | 36.25 (21.955) | 54.10 (28.276) | 66.42 (53.861)
  TGA peak, Change at Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  TGA peak, Change at Day 57 | 37.13 (21.866) | 32.57 (20.368) | 34.67 (20.584) | 33.93 (7.688) | 35.53 (15.716)
  TGA peak, Change at Day 85: number analyzed (Participants) | 7 | 5 | 6 | 6 | 13
  TGA peak, Change at Day 85 | 37.60 (21.142) | 69.92 (40.250) | 30.15 (18.614) | 30.15 (22.743) | 34.16 (21.306)
  TGA peak, Change at Day 113: number analyzed (Participants) | 7 | 2 | 4 | 6 | 13
  TGA peak, Change at Day 113 | 24.37 (33.703) | 16.05 (36.557) | 43.33 (68.794) | 6.93 (15.334) | 16.32 (27.345)

27. Secondary Outcome: Change From Baseline in Endogenous Thrombin Generation (TGA) Potential
Description: An ex vivo pharmacodynamic measure of thrombin generation. The endogenous TGA potential represents the total amount of active thrombin formed during thrombin generation and the peak height the maximal amount of thrombin formed.
Time Frame: Baseline, Study Day 2, 4, 8, 15, 22, 29, 30, 33, 57, 85 and 113
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: nanomole*minute
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
nanomole*minute
  Endogenous TGA Potential, Change at Day 2 | 864.0 (250.60) | 816.8 (211.13) | 999.8 (249.59) | 1065.3 (161.71) | 964.6 (227.95)
  Endogenous TGA Potential, Change at Day 4 | 766.7 (236.94) | 714.8 (275.75) | 808.7 (288.78) | 825.1 (294.44) | 795.9 (258.54)
  Endogenous TGA Potential, Change at Day 8 | 691.9 (301.43) | 659.8 (295.11) | 796.5 (151.00) | 918.6 (276.26) | 805.2 (301.66)
  Endogenous TGA Potential, Change at Day 15 | 674.9 (244.61) | 608.5 (242.81) | 800.8 (334.99) | 639.3 (145.74) | 657.1 (194.32)
  Endogenous TGA Potential, Change at Day 22 | 646.9 (295.05) | 589.0 (274.33) | 647.0 (236.38) | 731.4 (302.89) | 689.1 (290.60)
  Endogenous TGA Potential, Change at Day 29: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  Endogenous TGA Potential, Change at Day 29 | 588.2 (239.00) | 623.0 (188.84) | 618.3 (276.51) | 660.5 (340.36) | 624.3 (282.93)
  Endogenous TGA Potential, Change at Day 30: number analyzed (Participants) | 6 | 6 | 6 | 5 | 11
  Endogenous TGA Potential, Change at Day 30 | 494.8 (247.86) | 672.0 (226.25) | 603.3 (332.44) | 710.2 (272.54) | 592.7 (270.33)
  Endogenous TGA Potential, Change at Day 33: number analyzed (Participants) | 6 | 6 | 6 | 5 | 11
  Endogenous TGA Potential, Change at Day 33 | 716.5 (391.60) | 606.0 (280.39) | 583.7 (291.25) | 848.8 (387.17) | 776.6 (376.05)
  Endogenous TGA Potential, Change at Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  Endogenous TGA Potential, Change at Day 57 | 586.8 (200.04) | 445.2 (220.86) | 564.5 (287.43) | 579.7 (147.04) | 583.3 (167.42)
  Endogenous TGA Potential, Change at Day 85: number analyzed (Participants) | 7 | 5 | 6 | 6 | 13
  Endogenous TGA Potential, Change at Day 85 | 566.6 (202.22) | 812.2 (198.80) | 526.7 (297.03) | 493.7 (368.68) | 532.9 (280.20)
  Endogenous TGA Potential, Change at Day 113: number analyzed (Participants) | 7 | 2 | 4 | 6 | 13
  Endogenous TGA Potential, Change at Day 113 | 256.4 (347.91) | 50.5 (290.62) | 306.5 (440.04) | 142.3 (361.25) | 203.8 (344.10)

28. Secondary Outcome: Change From Baseline in Prothrombin Fragments 1 + 2
Description: An in vivo pharmacodynamic measure of thrombin generation (prothrombin cleavage). Prothrombin fragment 1+2 (F 1+2) is the amino terminus fragment of the prothrombin molecule. It is a polypeptide with a half-life of approximately 90 minutes. F 1+2 is released from prothrombin when prothrombin is converted to thrombin by the prothrombinase complex.
Time Frame: Baseline, Study Day 2, 4, 8, 15, 22, 29, 30, 33, 57, 85 and 113
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: picomole/liter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
picomole/liter
  Prothrombin fragments 1 + 2, Change at Day 2 | 430.0 (383.03) | 498.3 (484.40) | 275.7 (206.71) | 438.9 (507.68) | 434.4 (432.08)
  Prothrombin fragments 1 + 2, Change at Day 4 | 548.1 (455.67) | 1096.7 (1403.57) | 574.5 (363.37) | 730.3 (537.21) | 639.2 (487.82)
  Prothrombin fragments 1 + 2, Change at Day 8 | 450.3 (396.09) | 562.2 (605.07) | 413.0 (171.50) | 580.7 (259.63) | 515.5 (328.78)
  Prothrombin fragments 1 + 2, Change at Day 15 | 481.7 (330.26) | 349.7 (212.59) | 389.2 (228.56) | 571.1 (474.23) | 526.4 (395.34)
  Prothrombin fragments 1 + 2, Change at Day 22 | 608.1 (336.97) | 322.3 (161.76) | 420.2 (166.66) | 524.1 (577.08) | 566.1 (456.08)
  Prothrombin fragments 1 + 2, Change at Day 29: number analyzed (Participants) | 6 | 6 | 6 | 7 | 13
  Prothrombin fragments 1 + 2, Change at Day 29 | 650.3 (415.58) | 288.0 (259.19) | 577.7 (302.76) | 429.3 (257.91) | 531.3 (344.06)
  Prothrombin fragments 1 + 2, Change at Day 30: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  Prothrombin fragments 1 + 2, Change at Day 30 | 655.7 (496.35) | 486.0 (608.26) | 521.0 (165.25) | 580.8 (507.83) | 618.3 (480.35)
  Prothrombin fragments 1 + 2, Change at Day 33: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  Prothrombin fragments 1 + 2, Change at Day 33 | 761.3 (509.02) | 642.5 (759.02) | 1527.7 (2499.96) | 609.2 (380.74) | 685.3 (435.87)
  Prothrombin fragments 1 + 2, Change at Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  Prothrombin fragments 1 + 2, Change at Day 57 | 586.5 (473.53) | 216.5 (173.44) | 465.3 (300.84) | 463.5 (397.57) | 525.0 (421.78)
  Prothrombin fragments 1 + 2, Change at Day 85: number analyzed (Participants) | 7 | 5 | 6 | 6 | 13
  Prothrombin fragments 1 + 2, Change at Day 85 | 588.3 (483.80) | 378.2 (207.16) | 470.2 (244.21) | 362.2 (378.54) | 483.9 (436.47)
  Prothrombin fragments 1 + 2, Change at Day 113: number analyzed (Participants) | 7 | 2 | 4 | 6 | 13
  Prothrombin fragments 1 + 2, Change at Day 113 | -6.6 (151.87) | 16.5 (19.09) | -75.5 (76.86) | -58.2 (121.15) | -30.4 (135.52)

29. Secondary Outcome: Change From Baseline in D-Dimer
Description: An in vivo pharmacodynamic measure of thrombin generation (fibrin degradation). D-dimer is a fibrin degradation product, a small protein fragment present in the blood after a blood clot is degraded by fibrinolysis. D-dimer is one of the protein fragments produced when a blood clot gets dissolved in the body. It is normally undetectable or detectable at a very low level unless the body is forming and breaking down blood clots. Then, its level in the blood can significantly rise.
Time Frame: Baseline, Study Day 2, 4, 8, 15, 22, 29, 30, 33, 57, 85 and 113
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: microgram/milliliter
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
microgram/milliliter
  D-dimer, Change at Day 2 | 0.0393 (0.16303) | 0.0792 (0.22238) | 0.1900 (0.09301) | 0.1086 (0.30536) | 0.0739 (0.23790)
  D-dimer, Change at Day 4 | 0.2050 (0.24491) | 0.2842 (0.36896) | 0.3217 (0.23248) | 0.6729 (0.62524) | 0.4389 (0.51676)
  D-dimer, Change at Day 8 | 0.0743 (0.26111) | 0.2017 (0.29753) | 0.3292 (0.40635) | 0.5614 (0.54901) | 0.3179 (0.48422)
  D-dimer, Change at Day 15 | 0.0979 (0.25666) | 0.1942 (0.28748) | 0.2500 (0.23424) | 0.1900 (0.82310) | 0.1439 (0.58769)
  D-dimer, Change at Day 22 | 0.1364 (0.27802) | 0.2167 (0.33877) | 0.2000 (0.26109) | 0.1829 (1.27802) | 0.1596 (0.88887)
  D-dimer, Change at Day 29: number analyzed (Participants) | 6 | 6 | 6 | 7 | 13
  D-dimer, Change at Day 29 | 0.0633 (0.20029) | 0.2308 (0.32355) | 0.1517 (0.42347) | -0.0129 (1.17491) | 0.0223 (0.84172)
  D-dimer, Change at Day 30: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  D-dimer, Change at Day 30 | 0.1350 (0.32388) | 0.1492 (0.26345) | 0.2133 (0.33914) | -0.0833 (1.31549) | 0.0258 (0.92048)
  D-dimer, Change at Day 33: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  D-dimer, Change at Day 33 | 0.0800 (0.28796) | 0.1283 (0.37519) | 0.1233 (0.49855) | -0.1700 (1.68635) | -0.0450 (1.16076)
  D-dimer, Change at Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  D-dimer, Change at Day 57 | 0.1942 (0.30049) | 0.2175 (0.22554) | 0.1233 (0.36122) | 0.4033 (0.37120) | 0.2988 (0.34001)
  D-dimer, Change at Day 85: number analyzed (Participants) | 7 | 5 | 6 | 6 | 13
  D-dimer, Change at Day 85 | 0.1664 (0.30521) | 0.5860 (1.00003) | 0.1833 (0.43840) | 0.2300 (0.60395) | 0.1958 (0.44682)
  D-dimer, Change at Day 113: number analyzed (Participants) | 7 | 2 | 4 | 6 | 13
  D-dimer, Change at Day 113 | -0.1000 (0.22127) | 0.1875 (0.26517) | 0.0175 (0.41838) | -0.7833 (1.60090) | -0.4154 (1.10366)

30. Secondary Outcome: Change From Baseline in Dilute Prothrombin Time
Description: An ex vivo pharmacodynamic measure of thrombin generation (via extrinsic pathway). Clotting time is measured using a dilute prothrombin time reagent consisting of a unique formulation of relipidated recombinant tissue factor and calcium.
Time Frame: Baseline, Study Day 2, 4, 8, 15, 22, 29, 30, 33, 57, 85 and 113
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14
seconds
  Dilute prothrombin Time, Change at Day 2 | -27.84 (21.023) | -13.32 (25.780) | -31.25 (13.606) | -17.14 (26.167) | -22.49 (23.470)
  Dilute prothrombin Time, Change at Day 4 | -30.03 (24.312) | -17.87 (20.042) | -34.50 (18.306) | -14.70 (30.971) | -22.36 (27.907)
  Dilute prothrombin Time, Change at Day 8 | -23.63 (19.991) | -15.10 (22.129) | -31.23 (19.645) | -20.97 (33.969) | -22.30 (26.813)
  Dilute prothrombin Time, Change at Day 15 | -20.73 (23.070) | -19.33 (20.853) | -33.53 (14.880) | 1.11 (27.208) | -9.81 (26.753)
  Dilute prothrombin Time, Change at Day 22 | -21.40 (22.351) | -10.55 (16.057) | -26.78 (32.501) | -21.61 (30.842) | -21.51 (25.877)
  Dilute prothrombin Time, Change at Day 29: number analyzed (Participants) | 6 | 6 | 6 | 7 | 13
  Dilute prothrombin Time, Change at Day 29 | -15.32 (13.867) | -7.10 (20.643) | -40.40 (22.458) | -18.03 (24.600) | -16.78 (19.613)
  Dilute prothrombin Time, Change at Day 30: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  Dilute prothrombin Time, Change at Day 30 | -13.27 (13.399) | -23.45 (19.413) | -45.18 (21.372) | -17.47 (25.729) | -15.37 (19.680)
  Dilute prothrombin Time, Change at Day 33: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  Dilute prothrombin Time, Change at Day 33 | -23.35 (17.690) | -21.23 (20.010) | -29.10 (20.783) | -19.97 (19.297) | -21.66 (17.737)
  Dilute prothrombin Time, Change at Day 57: number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
  Dilute prothrombin Time, Change at Day 57 | -14.75 (14.393) | -12.03 (30.806) | -26.80 (12.911) | -11.72 (42.872) | -13.23 (30.531)
  Dilute prothrombin TIme, Change at Day 85: number analyzed (Participants) | 7 | 5 | 6 | 6 | 13
  Dilute prothrombin TIme, Change at Day 85 | -20.99 (25.424) | -25.80 (24.334) | -23.43 (26.166) | -12.42 (34.871) | -17.03 (29.148)
  Dilute prothrombin Time, Change at Day 113: number analyzed (Participants) | 7 | 2 | 4 | 6 | 13
  Dilute prothrombin Time, Change at Day 113 | -16.44 (13.578) | 14.30 (61.235) | -39.63 (20.182) | -12.78 (28.226) | -14.75 (20.682)

31. Secondary Outcome: Number of Participants Who Tested Positive for Anti-PF-06741086 Antibody (ADA)
Description: Human plasma ADA samples were analyzed for the detection of anti PF-06741086 antibodies by using semi-quantitative electrochemiluminescence (ECL) method. The criterion for positive result of ADA samples was ADA titer >=1.53. Treatment induced are negative prior to dosing and become positive during/after dosing. Treatment boosted are positive prior to dosing but titer increases during/after dosing.
Time Frame: Baseline up to Study Day 113
Population: This analysis population included all participants who received at least 1 dose of investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 7 | 6 | 6 | 7 | 14 | 26
Participants
  ADA incidence | 0 | 1 | 2 | 0 | 0 | 3
  Participants with treatment induced ADA incidence | 0 | 1 | 2 | 0 | 0 | 3
  Participants with treatment boosted ADA incidence | 0 | 0 | 0 | 0 | 0 | 0

32. Secondary Outcome: Number of Participants Who Tested Positive for Neutralizing Antibody (NAb)
Description: Human plasma NAb samples were analyzed for the presence or absence of NAb to PF-06741086 using semi-quantitative electrochemiluminescence (ECL) method. Treatment induced are negative prior to dosing and become positive during/after dosing. Treatment boosted are positive prior to dosing but titer increases during/after dosing.
Time Frame: Baseline up to Study Day 113
Population: Only positive ADA samples and the corresponding baseline sample were tested in the NAb assay.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
Number analyzed (Participants) | 0 | 1 | 2 | 0 | 0 | 3
Participants
  NAb incidence | 0 | 0 | 0 | 0 | 0 | 0
  Participants with treatment induced NAb incidence | 0 | 0 | 0 | 0 | 0 | 0
  Participants with treatment boosted NAb incidence | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 113 days
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | PF-06741086 300 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor | PF-06741086 450 mg SC QW Non-Inhibitor | PF-06741086 300 mg SC QW Inhibitor | Overall PF-06741086 300 mg SC | Total
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/7 | 0/14 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/6 | 1/6 | 1/7 | 2/14 | 4/26
Other Adverse Events (participants affected / at risk) | 6/7 | 4/6 | 6/6 | 4/7 | 10/14 | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06741086 300 mg SC QW Non-Inhibitor (N=7) | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor (N=6) | PF-06741086 450 mg SC QW Non-Inhibitor (N=6) | PF-06741086 300 mg SC QW Inhibitor (N=7) | Overall PF-06741086 300 mg SC (N=14) | Total (N=26)
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Physical assault (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-06741086 300 mg SC QW Non-Inhibitor (N=7) | PF-06741086 300 mg SC Loading + 150 mg SC QW Non-Inhibitor (N=6) | PF-06741086 450 mg SC QW Non-Inhibitor (N=6) | PF-06741086 300 mg SC QW Inhibitor (N=7) | Overall PF-06741086 300 mg SC (N=14) | Total (N=26)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Injection site bruising (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Injection site pain (General disorders) | 1 (2) | 1 (1) | 1 (6) | 0 (0) | 1 (2) | 3 (9)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 3 (4)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Occupational exposure to product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT02974855/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT02974855/SAP_001.pdf